CLINICAL TRIAL: NCT02217618
Title: A Single Dose Pharmacokinetic Study of LY2409021 Tablet Administered in Healthy Subjects
Brief Title: A Study of LY2409021 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14580; I1R-MC-GLDL (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — adomeglivant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2409021 (Experimental): Single oral dose of 20 milligrams (mg) LY2409021.
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: LY2409021

SUMMARY:
The study involves a single dose of LY2409021 taken by mouth. The purpose of this study is to determine how much LY2409021 enters the bloodstream and how long the body takes to get rid of the drug after the dose. This study will last approximately 28 days, not including screening. Screening can occur within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females as determined by medical history
* Satisfactory clinical laboratory and physical examination tests
* Have a body mass index (BMI) of 18 to 32.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

- Abnormal electrocardiograms (ECGs)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2409021
Started | 16
Received Study Drug | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- LY2409021: Single oral dose of 20 mg LY2409021.
Arm/Group | LY2409021
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2409021
Description: Area under the concentration versus time curve from zero to infinity (AUC[0-inf]) of LY2409021 is presented.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 144, 192, 264, and 336 hours post-dose
Population: All participants who received a dose of study drug and had evaluable AUC(0-inf) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliliter (ng*h/mL)
Arm/Group | LY2409021
Number analyzed (Participants) | 16
nanogram*hours per milliliter (ng*h/mL) | 48100 (28)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2409021
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 144, 192, 264, and 336 hours post-dose
Population: All participants who received a dose of study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2409021
Number analyzed (Participants) | 16
nanograms per milliliter (ng/mL) | 625 (29)

3. Primary Outcome: Pharmacokinetics: Time to Maximum Observed Drug Concentration (Tmax) of LY2409021
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 144, 192, 264, and 336 hours post-dose
Population: All participants who received a dose of study drug and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | LY2409021
Number analyzed (Participants) | 16
hours | 8.00 [4.00 to 24.03]

ADVERSE EVENTS:
Arm/Group | LY2409021
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days